CLINICAL TRIAL: NCT00474123
Title: Comparison of Antiplatelet and Anti-inflammatory Effects of High Dose Statin Monotherapy Versus Moderate Dose Statin Plus Ezetimibe
Brief Title: Antiplatelet and Anti-inflammatory Effects of Statins and Ezetimibe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: São Paulo Research Foundation (FAPESP), São Paulo Research Foundation (FAPESP)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 893/05
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Results first posted 2010-07-14 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-02

CONDITIONS: Stable Angina
Keywords: angina; atherosclerosis; simvastatin; ezetimibe; inflammation
MeSH Terms: conditions — Angina, Stable; Angina Pectoris; Atherosclerosis; Inflammation | interventions — Simvastatin; Ezetimibe; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin 80 mg (Active Comparator): Patients were treated with simvastatin 80 mg for 6 weeks
  Interventions: Drug: Simvastatin 80 mg/day for 6 weeks
- Ezetimibe 10 mg / Simvastatin 20 mg (Active Comparator): Patients were treated with daily Ezetimibe 10 mg / Simvastatin 20 mg for 6 weeks
  Interventions: Drug: Ezetimibe 10 mg / Simvastatin 20 mg

INTERVENTIONS:
Drug: Simvastatin 80 mg/day for 6 weeks — Simvastatin 80 mg/day, single dose, for 6 weeks.
  Other Names: Simvastatin 80 mg (Zocor)
  Arms: Simvastatin 80 mg
Drug: Ezetimibe 10 mg / Simvastatin 20 mg — Ezetimibe 10 mg / Simvastatin 20 mg
  Patients were treated with daily Ezetimibe 10 mg / Simvastatin 20 mg for 6 weeks
  Other Names: Vytorin
  Arms: Ezetimibe 10 mg / Simvastatin 20 mg

SUMMARY:
Among patients with stable coronary artery disease (CAD), it is not clear if the pleiotropic effects of cholesterol reduction differ between high-dose simvastatin alone and combined ezetimibe/simvastatin.

The investigators sought to compare the anti-inflammatory and anti-platelet effects of ezetimibe 10 mg / simvastatin 20 mg (E10/S20) to simvastatin 80 mg (S80).

DETAILED DESCRIPTION:
Introduction

Among patients with coronary artery disease (CAD), a robust evidence base supports the beneficial effects of statin therapy on mortality and other adverse cardiovascular outcomes . Recently, two large trials , have demonstrated that compared to standard dose statin therapy, high statin doses reduced Low-density lipoprotein-C (LDL-C) to extremely low levels and decreased coronary events, even in patients with normal levels of Low-density lipoprotein-C (LDL-C). Subsequently, recent guidelines have suggested an Low-density lipoprotein-C (LDL-C) treatment goal of <70 mg/dL in patients with coronary artery disease (CAD). Achieving such low Low-density lipoprotein-C (LDL-C) levels frequently demands an intensive Low-density lipoprotein-C (LDL-C) reduction, often above 50%. Ezetimibe, an intestinal cholesterol absorption inhibitor, can be used as an additional therapy if statin monotherapy fails to reduce Low-density lipoprotein-C (LDL-C) below the treatment goal.

Furthermore, anti-inflammatory and antithrombotic pleiotropic effects of statins might explain, at least in part, the large benefits demonstrated in randomized trials , . For example, in hypercholesterolemic patients treated with statins, a decrease in inflammation-associated markers such as the C-reactive protein (CRP) has been described , although it is debated whether this effect is clearly independent of Low-density lipoprotein-C (LDL-C).

Moreover, although inhibition of platelets by statin therapy is a well established effect , , it has not yet been clarified whether platelet inhibition by statin therapy depends on the reduction of Low-density lipoprotein-C (LDL-C) or on the inhibition of intracellular signal pathways accompanied by disaggregating effects.

Two alternative pharmacologic strategies are equally effective in reducing Low-density lipoprotein-C (LDL-C): high-dose statin alone and combined treatment with ezetimibe plus moderate-dose statin . It is not known whether these two strategies have different cholesterol-independent pleiotropic effects on inflammation and platelets. We therefore compared the anti-inflammatory and antiplatelet effects of two intensive pharmacologic strategies to reduce cholesterol: 80 mg of simvastatin (S80) versus 10 mg ezetimibe/ 20 mg of simvastatin (E10/S20). Anti-inflammatory effects were assessed by performing serial measurements of the following biomarkers: C-Reactive Protein (CRP), monocyte chemoattractant protein (MCP)-1, oxidized Low-density lipoprotein-C (oxLDL), soluble intercellular adhesion molecule (sICAM)-1. Platelet aggregation was also compared between the two strategies.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina
* Low-density lipoprotein (LDL) cholesterol 70-160 mg/dl

Exclusion Criteria:

* Renal failure
* Age>80
* Simvastatin current treatment>20mg
* Hepatic disease
* Inflammatory diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CARLOS V SERRANO, PHD, Principal Investigator — Heart Institute (InCor) HOSPITAL DAS CLINICAS DA FACULDADE DE MEDICINA DA UNIVERSIDADE DE SAO PAULO (HCFMUSP)
Locations (1):
- Heart Institute (InCor) HOSPITAL DAS CLINICAS DA FACULDADE DE MEDICINA DA UNIVERSIDADE DE SAO PAULO (HCFMUSP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Pesaro AE, Serrano CV Jr, Katz M, Marti L, Fernandes JL, Parra PR, Campos AH. Increasing doses of simvastatin versus combined ezetimibe/simvastatin: effect on circulating endothelial progenitor cells. J Cardiovasc Pharmacol Ther. 2013 Sep;18(5):447-52. doi: 10.1177/1074248413489771. Epub 2013 Jun 5. PMID 23739650
- [Derived] Pesaro AE, Serrano CV Jr, Katz M, Campos AH, Lopes RD, Marti LC, Martins HS, Sunahara RS, Maranhao RC, Nicolau JC. Inflammation and circulating endothelial progenitor cells in patients with coronary artery disease and residual platelet reactivity. Clinics (Sao Paulo). 2012 Sep;67(9):1117-21. doi: 10.6061/clinics/2012(09)21. No abstract available. PMID 23018312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2006 to January 2009, we randomized 78 patients with stable coronary artery disease (CAD) with LDL-C > 70 mg/dl, Angiographically documented CAD, stable angina, and age between 18 and 80 years. Patients were assigned randomly to two groups. The one group received Ezetimibe 10 mg/Simvastatin 20 mg the one other received Simvastatin 80 mg.
Pre-assignment Details: No wash-out period.
Groups:
- Simvastatin 20mg/Ezetimibe 10 mg: Patients were treated with Simvastatin 20mg/Ezetimibe 10 mgfor 6 weeks
Period: Overall Study
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Started | 38 | 40
Completed | 38 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 37 | 72
  >=65 years | 3 | 3 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10) | 64.5 (9) | 63.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 20 | 25 | 45
Region of Enrollment [Number; unit: participants]
  Brazil | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: C-reactive Protein
Description: Serum was separated by centrifugation from the blood samples. For high-sensitivity C-Reactive Protein measurement, whole venous blood was collected in tubes without anticoagulant and centrifuged at room temperature. Serum C-Reactive Protein was assessed with a high-sensitivity, latex microparticle-enhanced immunoturbidimetric assay (Behring Nephelometer Analyzer System; Behring Diagnostics, Somerville, NJ).
Time Frame: Change from baseline at 6 weeks
Population: per protocol
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
Percentage | -16 [-42 to 7] | -11 [-37 to 26]
Statistical Analysis 1: Comparison: Simvastatin 80 mg vs Simvastatin 20mg/Ezetimibe 10 mg; The sample size was determined as 78 patients. Continuous data were presented as means ± SD, or median (interquartile range) when the distribution was non-normal. For qualitative variables, we presented counts and relative frequencies. For between-group comparison we used multiple regression with adjustment for baseline values of the outcome variable (ANCOVA), or Wilcoxon rank-sum test when the variable had a non-normal distribution; Test type: Superiority or Other; p = 0.3, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Oxidized Low-Density Lipoprotein Cholesterol
Description: Serum samples were stored at -70°C and were determined simultaneously by ELISA in order to avoid variation of assay conditions. Commercial ELISA assays detecting oxLDL (Mercodia, USA) were applied.
Time Frame: Change from baseline at 6 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
Percentage | -18 (47) | -15 (33)
Statistical Analysis 1: Comparison: Simvastatin 80 mg vs Simvastatin 20mg/Ezetimibe 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.65, ANCOVA

3. Primary Outcome: Platelet Function Analyzer [PFA]-100
Description: Samples were collected in 3.8% sodium citrate (buffered, pH 5.5, Vacutainer, Becton Dickinson, Plymouth, UK) for platelet function tests. Platelet function assays were processed within 2 hours of blood collection. The PFA-100 records the closure time (CT), witch means the time in seconds (s) from the start of the test until the platelet plug occludes the aperture.
Time Frame: Change from baseline at 6 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
Percentage | 27 (43) | 8 (33)
Statistical Analysis 1: Comparison: Simvastatin 80 mg vs Simvastatin 20mg/Ezetimibe 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.02, ANCOVA

4. Primary Outcome: Monocyte Chemoattractant Protein (MCP)-1
Description: Serum samples were stored at -70°C and were determined simultaneously by ELISA in order to avoid variation of assay conditions. Commercial ELISA assays detecting MCP-1/ICAM-1 (R&D Systems, Europe, Abingdon, UK).
Time Frame: Change from baseline at 6 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
percentage | 11 (47) | 10 (21)
Statistical Analysis 1: Comparison: Simvastatin 80 mg vs Simvastatin 20mg/Ezetimibe 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.85, ANCOVA

5. Primary Outcome: Soluble Intercellular Adhesion Molecule (sICAM)-1
Description: as for outcome 4
Time Frame: Change from baseline at 6 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
percentage | 10 (14) | 10 (16)

6. Primary Outcome: Soluble CD40 Ligand
Description: A commercial ELISA assay detecting sCD40L (R&D Systems, USA) was applied. Detection limits and intra-assay variability was respectively, as follows: sCD-40L 15.6 pg/mL (intra-assay variability not available).
Time Frame: Fasting venous blood samples were drawn immediately after randomization and after at the conclusions of the six weeks study period.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
percentage | 6 (43) | 6 (34)

7. Primary Outcome: Interleukin-6
Description: A commercial ELISA assay detecting IL-6 (Siemens, USA) was applied.
Time Frame: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
percentage | 0 [-22 to 24] | 0 [-14 to 0]

8. Secondary Outcome: LDL Cholesterol
Time Frame: Fasting venous blood samples were drawn immediately after randomization and at the conclusions of the six week study period.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
percentage | -28 (30) | -29 (13)

9. Secondary Outcome: Triglyceride
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
percentage | -4 (32) | -14 (31)

10. Secondary Outcome: Endothelial Progenitor Cells
Description: Endothelial progenitor cells were evaluated by flow cytometry. Selected cells were positive for CD31, CD34 and VEGFR receptors.
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Number analyzed (Participants) | 38 | 40
percentage | 0.4 (1.7) | 0.1 (2.1)

ADVERSE EVENTS:
Arm/Group | Simvastatin 80 mg | Simvastatin 20mg/Ezetimibe 10 mg
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

LIMITATIONS AND CAVEATS:
Adverse Events were assessed, but none were observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes